CLINICAL TRIAL: NCT02967978
Title: Study on the Predictive Value of the Natural Calcium Isotope Ratio in Urine and Serum for the Diagnosis of Osteoporosis
Status: Completed | Type: Observational
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Dr. Christiane Laue, MD, Dr. med (medical doctor), Clinical Research Center Kiel GmbH
Other Study IDs: GEO-Osteo-2016
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Osteoporosis
Keywords: risk factors; Calcium isotopes; calcium turnover; DXA
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample, plasma sample, urine sample, stool sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims at investigating whether the natural calcium isotope ratio (δ44/40Ca) in urine and serum differs between postmenopausal women aged 50 to 75 years suffering from osteoporosis and a healthy control group and whether δ44/40Ca in urine and serum can be used for the diagnosis of osteoporosis or whether further parameters have to be included.

DETAILED DESCRIPTION:
According to the operational definition of WHO in the year 1994 osteoporosis is present if bone mineral content as assessed by DXA densitometry of the lumbar spine and/or proximal femur (total area or femoral neck) deviates from the mean of a 20 to 29 years old women by at least -2.5 standard deviations (DXA T-Score ≤ -2.5). This definition of osteoporosis is only valid after exclusion of other disorders, which may be associated with a reduction of bone mineral content and exclusion of osteomalacia.

By an individual screening 100 women will be included in the study who are characterized concerning existing or non-existing osteoporosis according to the guidelines of DVO 2014 and ISCD 2015, respectively.

According to the EPOS study results the prevalence of osteoporosis in Germany in postmenopausal women aged 50 to 60 years is about 15% and at the age of more than 70 years about 45%. In case of risk factors, such as hip fracture of father and/or mother, smoking, lactose intolerance, vegan nutrition, underweight (BMI < 20), diabetes, intake of loop diuretics, glucocorticoids, aromatase inhibitors and proton pump inhibitors a higher prevalence can be assumed. Thus by electing women with at least one risk factor of osteoporosis a higher proportion may meet the criteria of osteoporosis.

Since some women are expected to present with low vitamin D levels and so far are expected to present with osteomalacia, and since other exclusion criteria may occur, N = 100 women will be investigated, in order to obtain data from N = 80 women who may meet the criteria of the target group (about N = 40 with osteoporosis and about N = 40 without osteoporosis (normal control).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Age 50 - 75 years
* Fullfilling the criteria for diagnostic examination for osteoporosis incl. DXA according to DVO/ZÄS list 2015
* Written informed consent

Exclusion Criteria:

* known fracture within the last 3 months
* DXA within the last 12 month before inclusion
* Substitution with sex hormones
* Substitution with non-identified calcium supplements
* Vitamin D deficiency (post-hoc stratifying and exclusion from primary analysis, respectively)
* Hyperparathyreoidism (by history and based on calcium, phosphate and chloride in serum
* known renal failure
* known cancer disease
* Current enrollement in a clinical intervention trial
* Enrollement in a clinical intervention trial within the last 4 weeks
* Severe cognitive or psychiatric disorder
* Scheduled hospitalisation before the radiological examination (DXA)
* Legal incapacity

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 postmenopausal women aged 50- 75y having a risk for osteoporosis should be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
calcium isotope ratio δ44/40Ca in urine | 24 hours
  δ44/40Ca in urine of postmenopausal women who fulfill the criteria of osteoporosis are compared with δ44/40Ca in urine of those who do not fulfill the criteria using Mann-Whitney tests.

SECONDARY OUTCOMES:
the natural calcium isotope ratio δ44/40Ca in urine and serum (δ44/40Ca urine x serum) | 24 hours
  Elucidating whether the natural calcium isotope ratio δ44/40Ca in urine and serum (δ44/40Caurine x serum) differ between women with and without osteoporosis. For this purpose the δ44/40Caurine x serum of women who fulfill the criteria of osteoporosis are compared with δ44/40Caurine x serum of those who do not fulfill the criteria using Mann-Whitney tests.
turnover rate of calcium | 24 hours
  Elucidating whether the turnover rate of calcium in the total study population assessed by the existing compartment model correlates with markers of bone formation and bone resorption (P1NP x CTX).
  The level of significance will be adjusted for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, Dr. med, Principal Investigator — Clinical Research Center Kiel GmbH
Locations (1):
- Clinical Research Center Kiel GmbH, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No